CLINICAL TRIAL: NCT03896087
Title: Multicentre Clinical Trial to Assess the Performance of Centralized Assays for Hepatitis C Virus RNA Detection From Dried Blood Spot (DBS) Samples
Brief Title: Evaluation of Dried Blood Spot for HCV RNA Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 8160-2/1
Record Dates: First submitted 2019-03-14; First posted 2019-03-29 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hepatitis C, Chronic
Keywords: dried blood spots; plasma separation card; HCV RNA test
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clinical performance of the HCV DBS assay (Experimental): The study will be conducted in different geographical regions and populations and is designed to meet requirements of the for assays (medical devices) used for the qualitative and quantitative detection of Hepatitis C RNA.
  Interventions: Diagnostic Test: Abbott RealTime HCV assay from DBS; Diagnostic Test: HCV for use on the cobas® 6800/8800 Systems from PSC and DBS; Diagnostic Test: Aptima® HCV Quant Dx Assay from DBS; Diagnostic Test: HCV for use on the cobas® 4800Systems from PSC and DBS
- comparison PQ marked reference assay arm (Active Comparator): Plasma specimens from the participants will be tested on Abbott RealTime HCV assay that is approved for HCV diagnostics use by countries' authorities.
  Interventions: Diagnostic Test: Abbott RealTime HCV assay from DBS; Diagnostic Test: HCV for use on the cobas® 6800/8800 Systems from PSC and DBS; Diagnostic Test: Aptima® HCV Quant Dx Assay from DBS; Diagnostic Test: HCV for use on the cobas® 4800Systems from PSC and DBS

INTERVENTIONS:
Diagnostic Test: Abbott RealTime HCV assay from DBS — The trial intervention will consist of testing DBS, PSC and plasma samples obtained from trial participants using the centralised molecular assays for detection of HCV RNA. Results of testing DBS samples on the HCV assay will not be used to make any clinical decisions, and should not be communicated to study participants.
Diagnostic Test: HCV for use on the cobas® 6800/8800 Systems from PSC and DBS — The trial intervention will consist of testing DBS, PSC and plasma samples obtained from trial participants using the centralised molecular assays cobas® 6800/8800 Systems for detection of HCV RNA. Results of testing DBS samples on the HCV assay will not be used to make any clinical decisions, and should not be communicated to study participants.
Diagnostic Test: Aptima® HCV Quant Dx Assay from DBS — The trial intervention will consist of testing DBS, PSC and plasma samples obtained from trial participants using the centralised molecular assays Aptima® HCV Quant Dx Assay from DBS for detection of HCV RNA. Results of testing DBS samples on the HCV assay will not be used to make any clinical decisions, and should not be communicated to study participants.
Diagnostic Test: HCV for use on the cobas® 4800Systems from PSC and DBS — The trial intervention will consist of testing DBS, PSC and plasma samples obtained from trial participants using the centralised molecular assays cobas® 4800 for detection of HCV RNA. Results of testing DBS samples on the HCV assay will not be used to make any clinical decisions, and should not be communicated to study participants.

SUMMARY:
FIND is preparing a study to evaluate the performance, as measured by sensitivity and specificity, of four centralized assays for the detection of HCV RNA using capillary blood collected on dried blood spots (DBS) and plasma separation card (PSC).

DETAILED DESCRIPTION:
Available data on the performance of HCV RNA assays from DBS samples are insufficient to introduce their use in clinical practice. Only a few studies have been performed on DBS stored at ambient temperature, while the majority had DBS samples refrigerated or frozen right after collection, which does not mimic real-life settings. Additionally, due to the lack of standardized procedures, DBS collection and elution protocols varied across different studies. A large multicentre diagnostic accuracy study using standardized DBS collection and elution protocols validated by test manufacturers is needed to inform national hepatitis programmes and international guideline development groups. Test manufacturers need clinical evaluation data to update their regulatory claims and include DBS as an alternative sample type.

FIND is preparing a trial to evaluate the performance, as measured by sensitivity and specificity, of four laboratory-based assays for detection of HCV RNA assays using capillary blood collected on DBS/PSC. This will be provisional on the manufacturers agreeing to participate, as well as committing to applying to stringent regulatory approval for DBS/PSC.

ELIGIBILITY:
Three different population groups will be considered:

1. Individuals at risk of having HCV infection based on positive HCV serology test results

   Inclusion criteria:
   * Aged 18 years or older
   * Able to understand the scope of the trial
   * Provided written informed consent
   * Documented positive result of HCV serology test
2. Individuals at risk of having HCV infection based on past and/or current exposure to risk factors

   Inclusion criteria:
   * Aged 18 years or older
   * Able to understand the scope of the trial
   * Provided written informed consent
   * Past and/or current exposure to one of the high risk factors as defined by WHO and CDC guidelines (Appendix I)
3. Individuals diagnosed with chronic HCV infection who initiated or completed the anti-HCV treatment with direct acting antivirals (DAA) presenting at the clinical site for treatment monitoring or test of cure (i.e. sustained virological response)

Inclusion criteria:

* Aged 18 years or older
* Able to understand the scope of the trial
* Provided written informed consent
* Initiated on DAA treatment (regardless of type of DAA regimen) within 12 months prior to the enrolment to the trial

Exclusion criteria (for all trial populations):

* Previously enrolled in the trial
* Unwilling to provide required volume of fingerstick blood
* Unwilling to provide required volume of venous whole blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 942 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Point estimates (with 95% confidence intervals) of sensitivity and specificity for each assay for HCV RNA detection from DBS and/or PSC specimens measured against Abbott RealTime HCV VL assay performed at the clinical site | day 1 - day 30
  Point estimates (with 95% confidence intervals) of sensitivity and specificity for each assay for HCV RNA detection from DBS and/or PSC specimens measured against Abbott RealTime HCV VL assay performed at the clinical site
Evaluation of the correlation of HCV viral load level determined by each assay performed from DBS and/or PSC specimens with the HCV viral load level in plasma determined by Abbott RealTime HCV VL assay performed at the clinical site | day 1 - day 30
  Evaluation of the correlation of HCV viral load level determined by each assay performed

SECONDARY OUTCOMES:
Point estimates (with 95% confidence intervals) of sensitivity and specificity for each assay for HCV RNA detection from DBS and/or PSC specimens measured against the performance of the same assay in plasma | day 1 - day 30
  Point estimates (with 95% confidence intervals) of sensitivity and specificity for each assay for HCV RNA detection from DBS and/or PSC specimens measured against the performance of the same assay in plasma
Evaluation of the correlation of HCV viral load level determined by each assay performed from DBS and/or PSC specimens with the HCV RNA level in plasma determined by the same assay | day 1 - day 30
  Evaluation of the correlation of HCV viral load level determined by each assay performed from DBS and/or PSC specimens with the HCV RNA level in plasma determined by the same assay
WHO technician's appraisal sheet completed by all operators performing investigational test | through study completion, an average of 1 year
  WHO technician's appraisal sheet completed by all operators performing investigational test
point estimates (with 95% confidence intervals) of sensitivity and specificity for each assay for HCV RNA detection in plasma measured against the performance of Roche cobas® 6800 HCV VL assay | day 7 - day 30
  For Central Laboratory only
evaluation of the correlation of HCV RNA levels in plasma determined by each assay with HCV RNA levels in plasma determined by Roche cobas® 6800 HCV VL assay | day 7 - day 30
  For Central Laboratory only

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ivanova, Ph.D., Study Director — Foundation for Innovative New Diagnostics
Locations (5):
- St Vincent's Institute of Medical Research National Serology Reference Laboratory, Victoria Park, Fitzroy, Australia
- Centre Pasteur du Cameroun, Yaoundé, Yaounde, Cameroon
- National Centre for Disease Control, Tbilisi, Georgia
- Hellenic Scientific Society for the Study of AIDS and Sexually Transmitted Diseases, Athens, Greece
- Rwanda Military Hospital, Kigali, Kanombe, Rwanda

IPD SHARING:
Plan to Share IPD: No